CLINICAL TRIAL: NCT03110211
Title: Integration of Musculoskeletal Physical Therapy Care in the Patient Centered Medical Home
Acronym: IMPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Pro00081069
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-07

CONDITIONS: Musculoskeletal Pain Disorder
MeSH Terms: conditions — Collagen Diseases | interventions — Physicians, Primary Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapist Evaluation (Experimental): Patients are randomized to have an initial appointment with a physical therapist for a musculoskeletal complaint. The intervention is an initial evaluation and treatment recommendations by a physical therapist.
  Interventions: Procedure: Physical Therapist Evaluation
- Primary Care Physician Evaluation (Experimental): Patients are randomized to have an initial appointment with a primary care physician for a musculoskeletal complaint. The intervention is an initial evaluation and treatment recommendations by a primary care physician.
  Interventions: Procedure: Primary Care Physician

INTERVENTIONS:
Procedure: Physical Therapist Evaluation — Participants assigned to this group will receive an initial evaluation and treatment recommendations by a physical therapist.
  Other Names: PT First
  Arms: Physical Therapist Evaluation
Procedure: Primary Care Physician — Participants assigned to this group will receive an initial evaluation and treatment recommendations by a primary care physician.
  Other Names: PCP First
  Arms: Primary Care Physician Evaluation

SUMMARY:
Purpose and Objective: To determine the effectiveness of a physical therapist first versus a primary care physician first for patients entering a primary care setting with a musculoskeletal complaint on the outcomes of costs/charges, utilization and healthcare satisfaction.

Study activities and population group: This will be a randomized clinical trial enrolling patients who are seeking care to the Duke Outpatient Clinic with a musculoskeletal complaint. Patients, adults aged 18 years or greater, that agree to be part of the study will be randomized to see a physical therapist first or primary care physician first. All aspects of the evaluation and treatment by both providers will be standard care for musculoskeletal conditions.

Data analysis and risk/safety issues: Descriptive data including means and standard deviations and counts and proportions of baseline scores will be conducted. Differences in total costs/charges, opioid prescriptions, emergency department visits will be calculated and tested across groups. Participants may not personally be helped by taking part in this study. Participants may experience improvements in pain, function, or other symptoms from physical therapy program in this study. There is a minimal risk of loss of confidentiality. If a patient chooses not to participate, there will be no effect on their medical treatment and the study team will cease contact.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized clinical trial to examine the effectiveness an initial evaluation by a physical therapist compared to a primary care provider for patients with a musculoskeletal (MSK) complaint entering a primary care setting.

Background & Significance: MSK Conditions in Primary Care are Prevalent: More than 50% of the US population reported MSK conditions in 2011. The increase number of people over the age of 65 years will continue to increase the number of people with MSK conditions and increase demands on the health care system. The US healthcare system is already facing numerous challenges and care inefficiencies. Care for MSK conditions in primary care is an important area for care redesign to reduce inefficiencies. About 85% of people with MSK conditions have at least one visit with a primary care provider (PCP) and average six visits a year. Although, clinical guidelines recommend physical therapy as front-line care for MSK conditions, referrals to physical therapy for evaluation and management are disproportionate to the number in need. Uptake of these clinical guidelines is slow; yet advanced imaging and prescriptions for opioids for MSK pain is common. There was a 142% increase in the number of prescription medications filled by people with MSK conditions from 2009-2011. Overuse of opioids and advanced imaging and underuse of physical therapy can be deviated with novel care models that include physical therapists (PT) as frontline providers to where downstream healthcare utilization and costs are reduced and patients' needs are more directly met.

Coordinated care models can impact outcomes for prevalent conditions in primary care but data on MSK conditions is lacking: The high prevalence of depression among patients seeking primary care led to new models of integrated care. Co-location, for example, has proven successful for PCP and mental-health services, where it has almost doubled the rate of guideline based care, facilitating collaboration and referral due to proximity of specialized services. The current standard for primary care and patient-centered medical homes (PCMH) is for patients with MSK-related pain or complaints to be seen and evaluated by a PCP and then be recommended for advanced diagnostic imaging, opioids, or referral to PT at an offsite location (sometimes considered the medical neighborhood). Referral to an offsite location may negatively impact care continuity, provider communication and collaboration, and result in lower patient satisfaction from de-fragmented care and overuse of unnecessary services and prescription medication. Our approach to integrated and co-located PT could significantly decrease healthcare costs, improve patient satisfaction with care, decrease "no-show" PT rates and decrease physician burnout (by improving collaboration and satisfaction). In turn, changing mainstream MSK care.

Design & Procedures: This is a one-year randomized clinical trial of a novel health system redesign to study the immediate effect of a physical therapist first versus a primary care provider first for MSK conditions within a single primary care setting, the Duke Outpatient Clinic (DOC), at Duke University.

Randomization: This study will have two levels of randomization. Our biostatistician will generate the randomization schedule using a computerized random number generator with equal allocation to both groups for both levels of randomization. The investigators will use Redcap's Randomization Module to implement randomization scheme after consent to randomize appointments via phone. The first level consists of randomization to a Physical Therapist or Primary Care Physician as front line provider, both are considered standard of care approaches. The research coordinator will coordinate all randomization who will be blinded to the primary outcomes data collection. The second level of randomization will occur in the Primary Care Physician arm of the study. In this arm, if the Primary Care Physician decides physical therapy is medically necessary then the participant will be randomized to either be evaluated by an onsite Physical Therapist or receive a referral to be evaluated by an offsite Physical Therapist at a location of their choosing which is the current model of care at the DOC. This second level of randomization is so that the investigators can determine if physical therapy outcomes provided onsite are better when compared to offsite.

For participants that meet eligibility and following informed consent by the research coordinator, measures about demographics and health status will be completed. Patients assigned to the physical therapist first group will receive an evaluation by a licensed physical therapist onsite at the Duke Outpatient Clinic and be provided with a treatment plan of care for their MSK complaint(s). This evaluation and treatment plan of care will follow standard care currently implemented in clinical practice. Patients may return to the DOC for follow-up treatments if the physical therapist deems this treatment to be medically necessary. Patients assigned to the primary care provider group will receive an initial evaluation from a licensed primary care provider onsite. The evaluation by the primary care provider will follow standard care for evaluating MSK complaints in primary care. During the evaluation, the primary care provider may decide to refer to physical therapy or not for the patients with a MSK complaint. If the primary care provider refers to physical therapy the patient will be randomly assigned to either see the physical therapist onsite at the DOC or be assigned a referral to an offsite physical therapy clinic of the patients choosing with the assistance of the research coordinator. If the primary care provider decides that physical therapy is not medically necessary, the patient will follow the usual plan of care and treatment recommendations provided by their primary care provider. Following the visit, with either the physical therapist or primary care provider, the research coordinator will ask the patient to complete a short patient satisfaction survey about the initial visit. At approximately 3-months later the research coordinator will contact all enrolled patients by phone to collect health status questions and satisfaction with healthcare. Also, at 3-months outcomes related to total and MSK costs/charges will be collected by Duke University Health System Finance, outcomes of opioid prescriptions and emergency department visits during the 3-month period will be collected by electronic health record / administrative data (DEDUCE) and appointments to physical therapy that were referred offsite will be collect by administrative data from the Department of Physical Therapy / Occupational Therapy. The investigators will also collect, by electronic health record, usual care measures of functional status. The study will end following the 3-month follow-up phone call and outcomes and data are collected.

Study Interventions: All aspects related to physical therapy care are based on standard care provided by physical therapists for MSK complaints. Current practice at the Duke Outpatient Clinic consists of an onsite physical therapist to provide examinations, onsite exercise and home based exercise programs, and pain control education. Our planned study will consist of two interventions, both of which are standard care, however the investigators are modifying the order of when a patient may be seen by a physical therapist for a MSK complaint within the primary care setting. Our two interventions are physical therapist first or primary care provider first. The primary care provider first model may utilize the onsite physical therapist to provide physical therapy care by referral, known as the co-located primary care provider to physical therapist model, or utilize physical therapy by offsite referral.

Physical Therapist First. This model builds upon our current clinical model of a physical therapist co-located within the Duke Outpatient Clinic. This physical therapist has their own assigned treatment room, are known to the front desk scheduling staff for scheduling follow-up appointments, attend staff meetings and events and are considered a provider within the DOC system. Full support for their co-location is provided by the administration of the DOC and the Department of Physical and Occupational Therapy. The utilization of physical therapy services is considered standard care; however, the timing of services is unique given their co-location. This allows prompt access to not only physical therapy evaluation (billing for services occurs) but consultation with primary care provider (contact note for consultation in patients' medical records). For the current study, the investigators will utilize this already co-located physical therapist to be a front-line provider for musculoskeletal complaints of patients seeking care at the DOC. The physical therapist evaluation will be standard care for all patients seeking care to a physical therapist. It will not be modified in any way for the purposes of the study. If, at any time during evaluation the physical therapist determines that the patient would benefit from an additional primary care provider assessment, the patient will be scheduled for a primary care provider assessment, which may happen immediately following the physical therapist evaluation. In our experience these referrals from the physical therapist to primary care provider can occur within the same day, which adds considerable value to the efficiency of the integrated physical therapy model for those patients in need of additional primary care provider assessment.

Primary Care Provider First. In this model, patients would have an initial assessment from the primary care provider, which is considered standard care. If the primary care provider deems that the patient should be referred for physical therapy for medically necessary treatment, the research coordinator will randomly assign physical therapy referral to the onsite physical therapist at the Duke Outpatient Clinic or to an offsite location. The research coordinator will assist with scheduling and track referrals and all outcome data for patients referred offsite. In some cases, the primary care provider will not refer to physical therapy. In this case, the patients will follow the care recommendations provided by the primary care provider.

Data Analysis & Statistical Considerations: The investigators will calculate differences in total and MSK specific costs and charges between the physical therapist first group and the primary care provider group using standard T-tests or tests of medians depending on the distribution of data (parametric vs. non-parametric). The investigators will also calculate differences in the number of opioid prescriptions and emergency department visits between the two groups using chi-square categorical data analysis. The investigators will calculate changes in already routinely collected disease specific measures stored in electronic health record. Physical therapy missed appointments, patient and provider satisfaction will be reported as descriptive data. The investigators will also explore differences in outcomes of cost/charges, opioid prescriptions, emergency department visits and missed appointments between onsite provided physical therapy to offsite physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking care to the Duke Outpatient Clinic for a musculoskeletal complaint
* Patients speak English

Exclusion Criteria:

* Physical Therapist determines inappropriate for study due to medical reasons
* Patient does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Total patient costs accrued for musculoskeletal care during the 3 month study period | 3 months
  Total costs accrued for musculoskeletal care will be aggregated and abstracted by revenue code by the Duke University Health System Department of Finance
Total patient charges submitted for musculoskeletal care during the 3 month study period | 3 months
  Total charges submitted for musculoskeletal care will be aggregated and abstracted by revenue code by the Duke University Health System Department of Finance

SECONDARY OUTCOMES:
Patient Satisfaction with Healthcare | 3 months
  patient self reported satisfaction on the Patient Satisfaction Questionnaire (PSQ-8)
Opioid prescriptions | 3 months
  number of opioid prescriptions
Emergency Room Visits | 3 months
  number of emergency room visits
Imaging received | 3 months
  Number of imaging referrals received
Physical Therapy Missed Appointments | 3 months
  Number of missed appointments when referred from primary care physician to physical therapy clinic
Imaging Type | 3 months
  Type of imaging received
Provider Satisfaction | 3 months
  Primary care physician satisfaction will be measured with the Maslach Burnout Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Goode, DPT, PhD, Principal Investigator — Associate Professor
Locations (1):
- Duke Outpatient Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storheim K, Zwart JA. Musculoskeletal disorders and the Global Burden of Disease study. Ann Rheum Dis. 2014 Jun;73(6):949-50. doi: 10.1136/annrheumdis-2014-205327. No abstract available. PMID 24790065
- [Background] Goode AP, Freburger JK, Carey TS. The influence of rural versus urban residence on utilization and receipt of care for chronic low back pain. J Rural Health. 2013 Spring;29(2):205-14. doi: 10.1111/j.1748-0361.2012.00436.x. Epub 2012 Sep 27. PMID 23551651
- [Background] Carey TS, Freburger JK. Exercise and the Prevention of Low Back Pain: Ready for Implementation. JAMA Intern Med. 2016 Feb;176(2):208-9. doi: 10.1001/jamainternmed.2015.7636. No abstract available. PMID 26752108
- [Background] Freburger JK, Holmes GM, Agans RP, Jackman AM, Darter JD, Wallace AS, Castel LD, Kalsbeek WD, Carey TS. The rising prevalence of chronic low back pain. Arch Intern Med. 2009 Feb 9;169(3):251-8. doi: 10.1001/archinternmed.2008.543. PMID 19204216
- [Background] Carey TS, Freburger JK, Holmes GM, Castel L, Darter J, Agans R, Kalsbeek W, Jackman A. A long way to go: practice patterns and evidence in chronic low back pain care. Spine (Phila Pa 1976). 2009 Apr 1;34(7):718-24. doi: 10.1097/BRS.0b013e31819792b0. PMID 19282797
- [Background] Katon W. Health reform, research pave way for collaborative care for mental illness. Interview by Bridge M. Kuehn. JAMA. 2013 Jun 19;309(23):2425-6. doi: 10.1001/jama.2013.6494. No abstract available. PMID 23780435
- [Background] Woltmann E, Grogan-Kaylor A, Perron B, Georges H, Kilbourne AM, Bauer MS. Comparative effectiveness of collaborative chronic care models for mental health conditions across primary, specialty, and behavioral health care settings: systematic review and meta-analysis. Am J Psychiatry. 2012 Aug;169(8):790-804. doi: 10.1176/appi.ajp.2012.11111616. PMID 22772364
- [Derived] Carvalho E, Bettger JP, Bowlby L, Carvalho M, Dore D, Corcoran MW, Harris AA, Bond J, Goode AP. Integration of musculoskeletal physical therapy care in the patient-centred medical home (IMPaC): protocol for a single-site randomised clinical trial. BMJ Open. 2018 Aug 8;8(8):e022953. doi: 10.1136/bmjopen-2018-022953. PMID 30093522